CLINICAL TRIAL: NCT03072667
Title: Omegaven for Compassionate Use in the Treatment of Parenteral Nutrition-Associated Liver Disease
Status: Approved for marketing | Type: Expanded Access
Sponsor: Catherine Cibulskis, MD (Other)
Collaborators: St. Louis University (Other)
Responsible Party: Sponsor-Investigator, Catherine Cibulskis, MD, Assistant Professor of Pediatrics, St. Louis University
Organization: St. Louis University (Other)
Other Study IDs: 16150
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Cholestasis; Liver Diseases
Keywords: prematurity; bowel atresia; necrotizing entercolitis; parenteral nutrition associated liver disease (PNALD); intestinal failure; parenteral nutrition associated cholestasis; fish oil
MeSH Terms: conditions — Cholestasis; Liver Diseases; Premature Birth; Intestinal Atresia; Intestinal Failure | interventions — fish oil triglycerides

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Drug: Omegaven — Omegaven™ will be initiated at 0.5 gm fat/kg of body weight per day (5cc/kg per day of Omegaven™) for 2 days. On day 3, the rate of Omegaven™ will be increased to 1g/kg (10cc/kg) per day and will remain at this level thereafter unless otherwise indicated.

SUMMARY:
This is a compassionate use protocol of an investigational new drug (IND). The overall purpose of the treatment is to offer alternative treatment to children who developed parenteral nutrition-associated liver disease (PNALD) and have not responded positively to currently available medical therapies. PNALD develops in newborns dependent on parenteral nutrition (PN) and are unable to tolerate adequate enteral feedings to support fluid and nutritional fluids; although PN is necessary and life sustaining, it can result in severe liver disease.

DETAILED DESCRIPTION:
1. The overall purpose of the treatment is to offer alternative treatment to children who developed parenteral nutrition-associated liver disease (PNALD) and have not responded positively to currently available medical therapies. PNALD develops in newborns dependent on parenteral nutrition (PN) and are unable to tolerate adequate enteral feedings to support fluid and nutritional fluids; although PN is necessary and life sustaining, it can result in severe liver disease.

   The investigators want to see if a form of intravenous fat mixture, Omegaven, helps in the treatment of children with PNALD. Experimental data has shown that the intravenous fat mixture (Intralipid) that is currently being used as a part of newborn PN, may be contributing to the liver disease. Omegaven is different fat mixture manufactured and used in Europe in adults. It is different in that it is made from highly refined fish oil, while Intralipid is made from soybeans. Case control studies only, and not randomized clinical trials, show that Omegaven may reverse or treat PNALD. Since Omegaven is not currently approved for use in the United States, treatment IND was obtained from Food and Drug Administration (FDA).
2. Feeding intolerance is a common pathway of a broad array of medical and surgical disease states encountered in the neonatal population. Consequently, a high percentage of patients in neonatal intensive care units (NICU) need to rely on PN if they are to survive and grow. Through decades of research the development of PN has been a great success in that its use has maintained countless patients in sufficient nutritional status to recover from medical or surgical conditions. However, one complication of PN that remains poorly understood and that still causes considerable morbidity and mortality is PNALD.

   There are a wide variety of case scenarios for PNALD. There are scenarios in which newborns suffer irrecoverable bowel loss from some process (e.g., necrotizing enterocolitis totalis, mid gut volvulus) and consequently require long term PN as they await bowel transplant; as a result they almost always also require liver transplant secondary to PNALD. This further delays their surgery as they wait for two organs instead of one (Chungfat, Dixler et al. 2007). More commonly, cases involve patients who have prolonged bowel dysfunction that requires long term use of PN but who slowly recover and gradually transition to enteral feeds. For these infants the race between bowel recovery and PNALD progression often decides whether the patient lives or dies.
3. Although the etiology of PNALD is poorly understood and likely to be multi-factorial (Steinbach, Clark et al. 2008), recent animal research and human case studies suggest that altering the dose and the composition of the lipid component of PN might alter the course of PNALD (Alwayn, Gura et al. 2005; Gura, Parsons et al. 2005; Gura, Duggan et al. 2006; Gura, Lee et al. 2008). The lipid products used for PN in the United States are derived from soy oil; the brand used at Cardinal Glennon Children's Hospital is Intralipid®. Soy-based PN lipids are rich in omega-6 FA and also contain small amounts of omega-3 FA in the form of linolenic acid precursor. The potential toxicity of omega-6 fatty acids as it relates to PNALD has been recently revealed (Diamond, Sterescu et al. 2008; de Meijer, Gura et al 2009). This FA composition is sufficient to prevent essential FA deficiency (EFAD), historically measured as the ratio of specific omega-6 FA in the blood (Gura, Lee et al 2009).

In a published article (Gura, Duggan et al. 2006) reporting 2 cases in depth and in a subsequent paper (Gura, Lee et al. 2008) reporting 18 patients with established PNALD who required continued PN, investigators replaced the standard soy based lipid component of PN with a fish oil derived parenteral lipid (Omegaven™) that contains a high percentage (30 to 60%) of omega-3 FA. This therapy, which is still experimental in the United States, was associated with a gradual but ultimately profound correction of PNALD as indicated by laboratory markers such as conjugated bilirubin and circulating liver enzymes; the median time to reduce serum direct bilirubin from >2mg/dl to <2mg/dl was 9.4 weeks. No significant adverse effects of Omegaven™ in the doses utilized were identified.

The current study is to identify infants with PNALD of moderate severity or worse, defined as two consecutive measurements of direct bilirubin of 3 mg/dL after being on PN for > 3 weeks and who are anticipated to require PN for another 3 weeks, which puts them at risk of further progression of PNALD. For inclusion, other causes of liver disease must be ruled out. Upon meeting entry criteria, infant families will be offered, through an Institutional Review Board (IRB) approved consent process, the same treatment protocol for their infants that was successfully applied in the above cited clinical cases and detailed below. Monitoring for side effects, complications and disease progression or regression will be instituted. Therapy will be stopped when direct bilirubin is < 1 mg/dL for 2 weekly measurements or when the patient is tolerating enough enteral nutrition so that PN is no longer needed. Clinical and laboratory monitoring will be continued for 2 weeks post Omegaven™ infusion and as indicated by events thereafter. Additional endpoint criteria are: patients receiving transplants; AST/ALT, GGTP, C-reactive protein and albumin, mortality, infection rates and types, and frequency of red blood cell transfusions; if infant worsens with treatment or does not tolerate treatment with Omegaven, specifically for the adverse event of severe uncontrolled bleeding as listed in the risk section.

ELIGIBILITY:
Inclusion Criteria:

1. Age < 1 years; inpatient use only
2. PN dependency (unable to meet nutritional needs solely by enteral nutrition);
3. Present PNALD, as evidenced by two consecutive direct bilirubin > 3.0 mg/dL (at interval of one week);
4. Failed standard therapies to prevent the progression of liver disease:

   Avoiding overfeeding, reduction/removal of copper and manganese from PN, advancement of enteral feeding and the use of Ursodiol, if possible.
5. At the time the diagnosis PNALD is made, the patient is expected to continue PN at least an additional 3 weeks

Exclusion Criteria:

1. Any other cause of chronic liver disease (i.e., hepatitis B or C, cystic fibrosis, biliary atresia, or alpha 1 anti-trypsin deficiency etc.)
2. enrollment in any other clinical trial involving an investigational agent (unless approved by the designated physicians on the multidisciplinary team);
3. Lack of informed consent;
4. Intent to transfer to another healthcare facility
5. allergy to any seafood product, egg protein, and/or previous allergy to Omegaven
6. active coagulopathy characterized by ongoing bleeding or by a requirement for clotting factor replacement (e.g. fresh frozen plasma or cryoprecipitate) to maintain homeostasis
7. impaired lipid metabolism or severe hyperlipidemia with or without pancreatitis
8. unstable DM or hyperglycemia
9. stroke/embolism
10. collapse and shock
11. undefined coma status
12. recent MI
13. cholestasis due to any reason other than PNALD
14. active new infection at time of initiation of Omegaven
15. hemodynamic instability
16. unable to tolerate necessary laboratory monitoring
17. severe renal insufficiency

Max Age: 1 Year | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Locations (1):
- SSM Health Cardinal Glennon Children's Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Steinbach M, Clark RH, Kelleher AS, Flores C, White R, Chace DH, Spitzer AR; Pediatrix Amino-Acid Study Group. Demographic and nutritional factors associated with prolonged cholestatic jaundice in the premature infant. J Perinatol. 2008 Feb;28(2):129-35. doi: 10.1038/sj.jp.7211889. Epub 2007 Dec 6. PMID 18059467
- [Background] Alwayn IP, Gura K, Nose V, Zausche B, Javid P, Garza J, Verbesey J, Voss S, Ollero M, Andersson C, Bistrian B, Folkman J, Puder M. Omega-3 fatty acid supplementation prevents hepatic steatosis in a murine model of nonalcoholic fatty liver disease. Pediatr Res. 2005 Mar;57(3):445-52. doi: 10.1203/01.PDR.0000153672.43030.75. Epub 2005 Jan 19. PMID 15659701
- [Background] Gura KM, Parsons SK, Bechard LJ, Henderson T, Dorsey M, Phipatanakul W, Duggan C, Puder M, Lenders C. Use of a fish oil-based lipid emulsion to treat essential fatty acid deficiency in a soy allergic patient receiving parenteral nutrition. Clin Nutr. 2005 Oct;24(5):839-47. doi: 10.1016/j.clnu.2005.05.020. PMID 16029913
- [Background] Gura KM, Duggan CP, Collier SB, Jennings RW, Folkman J, Bistrian BR, Puder M. Reversal of parenteral nutrition-associated liver disease in two infants with short bowel syndrome using parenteral fish oil: implications for future management. Pediatrics. 2006 Jul;118(1):e197-201. doi: 10.1542/peds.2005-2662. PMID 16818533
- [Background] Gura KM, Lee S, Valim C, Zhou J, Kim S, Modi BP, Arsenault DA, Strijbosch RA, Lopes S, Duggan C, Puder M. Safety and efficacy of a fish-oil-based fat emulsion in the treatment of parenteral nutrition-associated liver disease. Pediatrics. 2008 Mar;121(3):e678-86. doi: 10.1542/peds.2007-2248. PMID 18310188
- [Background] Diamond IR, Sterescu A, Pencharz PB, Wales PW. The rationale for the use of parenteral omega-3 lipids in children with short bowel syndrome and liver disease. Pediatr Surg Int. 2008 Jul;24(7):773-8. doi: 10.1007/s00383-008-2174-0. Epub 2008 May 27. PMID 18504595
- [Background] de Meijer VE, Gura KM, Le HD, Meisel JA, Puder M. Fish oil-based lipid emulsions prevent and reverse parenteral nutrition-associated liver disease: the Boston experience. JPEN J Parenter Enteral Nutr. 2009 Sep-Oct;33(5):541-7. doi: 10.1177/0148607109332773. Epub 2009 Jul 1. PMID 19571170
- [Background] Park HW, Lee NM, Kim JH, Kim KS, Kim SN. Parenteral fish oil-containing lipid emulsions may reverse parenteral nutrition-associated cholestasis in neonates: a systematic review and meta-analysis. J Nutr. 2015 Feb;145(2):277-83. doi: 10.3945/jn.114.204974. Epub 2014 Dec 17. PMID 25644348